CLINICAL TRIAL: NCT00922792
Title: An Open, Non-Randomised Single and Multiple Dose Trial Investigating the Safety and Pharmacokinetics of Intravenous Administration of Long Acting rFVIIa (LA-rFVIIa) in Patients With Haemophilia A and B
Brief Title: Safety and Mode of Action of a Single Dose and Multiple Doses of Long Acting Activated Recombinant Human Factor VII in Patients With Haemophilia A and B
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7128-3700; 2009-010080-16 (EudraCT Number)
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia B
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: activated recombinant human factor VII, long acting
- B (Experimental)
  Interventions: Drug: activated recombinant human factor VII, long acting

INTERVENTIONS:
Drug: activated recombinant human factor VII, long acting — Single dose of 0,2 mg/kg LA-rFVIIa injected i.v. (intravenous) of 2 minutes duration
  Arms: A
Drug: activated recombinant human factor VII, long acting — Multiple doses of 100 mg/kg LA-rFVIIa injected i.v. (intravenous) of 2 minutes duration every 48 hours
  Arms: B

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the safety and pharmacokinetics (the effect of the body on the investigated drug) of long acting activated recombinant human factor VII (LA-rFVIIa) in patients with haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Haemophilia A or B
* Bodyweight max 100 kg
* Body Mass Index (BMI) max 30 kg/m2
* Adequate venous access

Exclusion Criteria:

* Known or suspected allergy to trial product(s) or related products (including NovoSeven®)
* The receipt of any investigational product within 30 days prior to enrolment in this trial
* Receipt of Immune Tolerance Induction (ITI) within the last 1 month prior to participation in this trial
* The receipt of any haemostatic treatment for control of a bleeding episode within the last 5 days prior to administration of trial product
* Receipt of FVIII or FIX replacement therapy within 48 hours prior to trial product administration
* Known pseudo tumours
* Congenital or acquired coagulation disorders other than haemophilia A or B
* Any major and/or orthopaedic surgery within one month prior to trial start
* Advanced atherosclerotic disease (defined as known history of ischemic heart disease, ischemic stroke, etc.)
* Clinical signs of renal dysfunction
* Use of platelet inhibitors, including NSAIDs, one week prior to administration of trial drug
* Use of non-prescribed opiate substances

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events | after 1 and 2 weeks after dosing
Frequency of serious adverse events | after 1, 2 and 6-10 weeks after dosing
Frequency of MESIs (Medical Event of Special Interest) | after 1, 2 and 6-10 weeks after dosing
Frequency of ocurrence of neutralising antibodies against FVII and/or LA-rFVIIa | after 2 and 6-10 weeks after dosing

SECONDARY OUTCOMES:
Pharmacokinetic parameters based on FVIIa activity. The pharmacokinetic parameters to be reported are: AUC(0-48h), AUC(0-t) and AUC, C10min, Vz, CL, and t½ | from time of dosing up to 72 hours after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Madrid, Spain

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com